CLINICAL TRIAL: NCT01073436
Title: Discontinuation of Tyrosine Kinase Inhibitor Therapy in Patients With Chronic-Phase Chronic Myeloid Leukemia, Previously Treated With Interferon-Alpha
Brief Title: Discontinuation of Imatinib Mesylate in Patients With Chronic-Phase Chronic Myeloid Leukemia Previously Treated With Interferon-Alpha
Status: Terminated | Type: Observational
Why Stopped: Closed prematurely due to low accrual.
Sponsor: University of Michigan Rogel Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: UMCC 2008.083; HUM00021950 (Other: University of Michigan Medical IRB)
Record Dates: First submitted 2010-02-19; First posted 2010-02-23 (Estimated); Last update posted 2016-11-15 (Estimated); Status verified 2016-11

CONDITIONS: Chronic Myeloid Leukemia
Keywords: diagnosis of Ph+) CML in chronic phase.; prior therapy with interferon-alpha for at least 2 years, and achieved at least a partial cytogenetic response; receiving a TKI (imatinib mesylate, dasatinib, nilotinib); WBC ≤ 10 x 109/L.; Platelet count < 450,000 x 109/L.; No blasts or promyelocytes in peripheral blood.; No evidence of disease-related symptoms and extramedullary disease; complete cytogenetic response (CCyR) on a TKI for a minimum of 1 yr; major molecular remission on a TKI for a minimum of 1 yr; 18 years of age or older; ECOG performance status of 0-2 (Appendix 13.1); Informed Consent
MeSH Terms: conditions — Leukemia, Myelogenous, Chronic, BCR-ABL Positive

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Discontinuation: Subjects who agree to discontinue their tyrosine kinase inhibitor(TKI)therapy, namely,imatinib mesylate, dasatinib, or nilotinib,and then followed to see if they can maintain a durable remission.
  Interventions: Other: Discontinuation of therapy

INTERVENTIONS:
Other: Discontinuation of therapy — Patients with chronic-phase chronic myeloid leukemia (CP-CML) previously treated with interferon-alpha (IFN) and presently on a tyrosine kinase inhibitor (TKI) (imatinib mesylate, dasatinib, or nilotinib) with achievement of a complete cytogenetic and at least a major molecular remission.

SUMMARY:
To investigate whether patients with chronic-phase chronic myeloid leukemia (CP-CML) previously treated with interferon-alpha (IFN) and presently on a tyrosine kinase inhibitor (TKI) (imatinib mesylate, dasatinib, or nilotinib) with achievement of a complete cytogenetic and at least a major molecular remission, are able to discontinue therapy and maintain a durable remission. Relapse-free survival (RFS) rate at 1 year after discontinuation of TKI will be the measurement of this objective.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must have a diagnosis of Philadelphia chromosome positive (Ph+) chronic myeloid leukemia in chronic phase.
2. Patients must have received prior therapy with interferon-alpha for their CML, for a period of at least 2 years, and achieved at least a partial cytogenetic response on this therapy, defined as 1% - 34% Ph+ cells in metaphase, present in the bone marrow.
3. Patients must be actively receiving treatment for their CML with a TKI (imatinib mesylate, dasatinib, nilotinib). If patients are receiving dasatinib or nilotinib, this can only be for reasons other than imatinib-resistant CML.
4. Patients must have an ongoing complete hematologic response (CHR) on a TKI, defined as follows:

   * WBC ≤ 10 x 109/L.
   * Platelet count < 450,000 x 109/L.
   * No blasts or promyelocytes in peripheral blood.
   * No evidence of disease-related symptoms and extramedullary disease, including the liver and spleen.
5. Patients must have a complete cytogenetic response (CCyR) on a TKI for a minimum of one year leading up to enrollment. Complete cytogenetic response is defined as 0% Ph+ cells in metaphase, in the bone marrow and/or a negative peripheral blood FISH analysis for the BCR/ABL gene fusion, and an ongoing CCyR must be confirmed by bone marrow aspirate cytogenetics and/or peripheral blood FISH for BCR/ABL within 4 weeks of discontinuing therapy.
6. Patients must have at least a major molecular remission on a TKI for a minimum of 1 year, present on 2 consecutive analyses, performed at least 3 months apart, in the 6 to 12 months leading up to enrollment. Major molecular remission is defined as ≥ 3 log reduction from a standard baseline value (equivalent to a BCR-ABL/ABL of ≤ 0.1%) in BCR/ABL transcript by quantitative RT-PCR performed on peripheral blood or bone marrow aspirate. Complete molecular remission is defined as a negative quantitative RT-PCR (QPCR) analysis for BCR/ABL, present on 2 consecutive analyses, performed at least 3 months apart, in the 6 to 12 months leading up to enrollment.
7. Patients must be eighteen years of age or older
8. Patients must have an ECOG performance status of 0-2 (Appendix 13.1)
9. All patients must be informed of the investigational nature of this study and standard alternative therapy. All patients must sign and give written informed consent in accordance with institutional and federal guidelines.

Exclusion Criteria:

1. Patients who have had prior progression of their CML to accelerated phase or blast crisis.
2. Patients who have previously undergone hematopoietic stem cell transplantation.
3. Patients receiving dasatinib or nilotinib due to a prior history of imatinib-resistant CML.
4. Patients with a history of non-compliance to medical regimens or who are considered potentially unreliable.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Diagnosed with Philadelphia chromosome positive (Ph+) chronic myeloid leukemia in chronic phase.
Sampling Method: Non-Probability Sample
Enrollment: 7 (Actual)
Dates: Start 2009-05; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
Relapse-free survival | 1 year
  Relapse-free survival (RFS) rate at 1 year after discontinuation of TKI will be the measurement of this objective.

SECONDARY OUTCOMES:
Reduction of the malignant stem cell population | 1 Year
  To determine whether prior treatment with interferon-alpha followed by TKI therapy effectively depletes/reduces the malignant stem cell population in CP-CML.

CONTACTS AND LOCATIONS:
Overall Officials: Dale Bixby, M.D./PhD, Principal Investigator — University of Michigan Rogel Cancer Center
Locations (1):
- University of Michigan Cancer Center, Ann Arbor, Michigan, United States